CLINICAL TRIAL: NCT07065526
Title: The Effect of Emotional Freedom Technique Applied to Postmenopausal Women on Sleep and Quality of Life: A Randomized Controlled Study
Brief Title: Application of EFT in Postmenopausal Women
Acronym: Postmenopausal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Merve Yazar, PhD, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KTO Karatay University
Record Dates: First submitted 2024-11-12; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Postmenopausal; Sleep; Quality of Life
Keywords: quality of life; Emotional freedom technique; postmenopausal women; sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Emodin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EFT Group (Experimental): Following the pre-test in the first encounter, the participants were administered the first EFT lasting 30-40 minutes by the first author, who is a certified EFT facilitator, followed by the CPS. Afterwards, a total of 4 sessions of EFT were administered at 1-week intervals. The CPS was applied before and after each EFT. After the last EFT session, SUE, PSQI and MENQOL post-tests were administered.
  Interventions: Behavioral: Emodin
- Control group (No Intervention): Following the pre-test application, post-tests were applied 4 weeks later. They received routine treatment and care. The control group was taught EFT application after the study was completed.

INTERVENTIONS:
Behavioral: Emodin — Following the pre-test in the first encounter, the participants were administered the first EFT lasting 30-40 minutes by the first author, who is a certified EFT facilitator, followed by the CPS. Afterwards, a total of 4 sessions of EFT were administered at 1-week intervals. The CPS was applied before and after each EFT. After the last EFT session, SUE, PSQI and MENQOL post-tests were administered.
  Arms: EFT Group

SUMMARY:
Objectives: This study was conducted to determine the effect of emotional liberation technique on sleep and quality of life in postmenopausal women.

Methods: The study was conducted as a randomized controlled trial with 58 women in a university hospital in Turkey. Of the women, 29 were in the intervention group and 29 were in the control group. Data were collected using the Personal Information Form, Subjective Experience Unit Scale (SUE), Pittsburg Sleep Quality Index (PSQI) and Menopause Specific Quality of Life Scale (MENQOL). EFT was applied to women in the intervention group four times at one-week intervals. The emotional liberation technique was applied to the women in the control group after the post-test was applied and the data were reported.

ELIGIBILITY:
Inclusion Criteria:

* Between 45 and 60 years old,
* No menstruation for at least 12 months
* A score of 5 or higher on the Pittsburgh Sleep Quality Index (PSQI)
* Conscious postmenopausal women who can read and write Turkish and have person, place, and time orientation

Exclusion Criteria:

* Anyone with an intellectual disability or diagnosed psychiatric illness, anyone taking medications that may affect sleep patterns, anyone on hormone replacement therapy,
* People who have previously been trained in EFT and have communication problems.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Sleep quality | 1 Month Follow-up
  The emotional freedom technique was applied four times a week.These results are evaluated using the Pittsburgh Sleep Quality Index. A total scale score of 5 or above is considered poor sleep.The higher the score on the scale, the lower the sleep quality.

SECONDARY OUTCOMES:
Menopause-Specific Quality of Life | 1 Month Follow-up
  The emotional freedom technique was applied four times a week. These results were evaluated using the Menopause-Specific Quality of Life Questionnaire. The lowest possible score on the scale is 0 and the highest is 154. As the score on the scale increases, the severity of the symptoms increases and quality of life decreases.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - KTO Karatay University, Karatay, Konya
  - Necmettin Erbakan Üniveristesi Tıp Fakültesi Hastanesi, Konya, Meram

IPD SHARING:
Plan to Share IPD: No